CLINICAL TRIAL: NCT04034095
Title: The Registry to Observe Clinical Outcomes of Patients With High-risk Metastatic Hormone-naïve Prostate Cancer in Japan
Brief Title: A Registry Study to Observe Clinical Outcomes of Participants With High-risk Metastatic Hormone-naïve Prostate Cancer in Japan
Status: Completed | Type: Observational
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Other Study IDs: CR108675; 56021927PCR4009 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2019-07-16; First posted 2019-07-26 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Prostatic Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Androgen Antagonists; bicalutamide; abiraterone; Prednisolone; Docetaxel; enzalutamide; apalutamide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: ADT alone/ ADT + Bicalutamide: Participants with diagnosis of metastatic hormone-naive prostate cancer (mHNPC) receiving androgen-deprivation therapy (ADT) alone or ADT plus bicalutamide (combined androgen blockade [CAB]) under routine clinical practice will be observed.
  Interventions: Drug: Androgen-deprivation Therapy (ADT); Drug: Bicalutamide
- Cohort 2: ADT + AAP/Docetaxel/Enzalutamide/Apalutamide: Participants with diagnosis of mHNPC receiving ADT plus abiraterone plus prednisolone (AAP) or Docetaxel or Enzalutamide or Apalutamide under routine clinical practice will be observed.
  Interventions: Drug: Androgen-deprivation Therapy (ADT); Drug: Abiraterone; Drug: Prednisolone; Drug: Docetaxel; Drug: Enzalutamide; Drug: Apalutamide

INTERVENTIONS:
Drug: Androgen-deprivation Therapy (ADT) — Participants enrolled in this study will continue to receive ADT (example- Leuprorelin, Goserelin and Degarelix) alone or in combination with other therapies in routine clinical practice as directed by their treating physician. No intervention will be administered as a part of this study.
Drug: Bicalutamide — Participants enrolled in this study will continue to receive bicalutamide along with ADT in routine clinical practice as directed by their treating physician. No intervention will be administered as a part of this study.
  Groups: Cohort 1: ADT alone/ ADT + Bicalutamide
Drug: Abiraterone — Participants enrolled in this study will continue to receive abiraterone in combination with prednisolone along with ADT in routine clinical practice as directed by their treating physician. No intervention will be administered as a part of this study.
  Groups: Cohort 2: ADT + AAP/Docetaxel/Enzalutamide/Apalutamide
Drug: Prednisolone — Participants enrolled in this study will continue to receive prednisolone in combination with abiraterone along with ADT in routine clinical practice as directed by their treating physician. No intervention will be administered as a part of this study.
  Groups: Cohort 2: ADT + AAP/Docetaxel/Enzalutamide/Apalutamide
Drug: Docetaxel — Participants enrolled in this study will continue to receive docetaxel along with ADT in routine clinical practice as directed by their treating physician. No intervention will be administered as a part of this study.
  Groups: Cohort 2: ADT + AAP/Docetaxel/Enzalutamide/Apalutamide
Drug: Enzalutamide — Participants enrolled in this study will continue to receive enzalutamide along with ADT in routine clinical practice as directed by their treating physician. No intervention will be administered as a part of this study.
  Groups: Cohort 2: ADT + AAP/Docetaxel/Enzalutamide/Apalutamide
Drug: Apalutamide — Participants enrolled in this study will continue to receive apalutamide along with ADT in routine clinical practice as directed by their treating physician. No intervention will be administered as a part of this study.
  Groups: Cohort 2: ADT + AAP/Docetaxel/Enzalutamide/Apalutamide

SUMMARY:
The purpose of this registry study is to longitudinally observe clinical outcomes and patient-reported outcomes (PRO) for participants with high-risk metastatic hormone-naive prostate cancer (mHNPC) in the real-world setting in Japan.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of metastatic, hormone-naïve prostate cancer (mHNPC) after 1 May 2019
* Should have at least 2 of the 3 following high-risk factors: a Gleason score of greater than or equal to (>=) 8, at least 3-bone lesions, or the presence of visceral metastasis
* Willing to receive androgen-deprivation therapy (ADT) containing regimens for high-risk metastatic, hormone-naïve prostate cancer (mHNPC) in the hospital which have the contract with sponsor for this study, or patient received a regimen containing ADT for high-risk mHNPC
* Possess Japanese nationality
* Each patient (or their legally acceptable representative) must sign an informed consent form (ICF) indicating that he understands the purpose of, and procedures required for the study and is willing to participate in the study. For dead cases, the ICF can be waived after approved by Independent Ethics Committee/Institutional Review Board (IEC/IRB)

Exclusion Criteria:

- has any other active malignancies

Min Age: 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with high-risk metastatic hormone-naive prostate cancer (mHNPC) in Japan receiving androgen-deprivation therapy (ADT) containing treatment under routine clinical practice will be observed throughout their course of treatment, during which data on prostate cancer (PC) treatment, radiographic/clinical progression, and outcomes (including death) will be collected. The main source of data collection will be medical records of each participating participant.
Sampling Method: Non-Probability Sample
Enrollment: 979 (Actual)
Dates: Start 2019-07-08 (Actual); Primary Completion 2024-08-13 (Actual); Study Completion 2024-08-13 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants who Achieve Prostate-specific Antigen (PSA) <=0.2 ng/mL Within a Year from Registration | 1 year
  Percentage of participants who achieve prostate-specific antigen (PSA) less than or equal to (<=)0.2 nanogram per milliliter (ng/mL) within a year from registration will be reported.
PSA Progression-free Survival (PSA-PFS) | Up to 5 years
  The PSA-PFS is defined as the duration from registration to either PSA progression or death, whichever occurs first.
Percentage of Participants with PSA-PFS | 2 years
  Percentage of participants with PSA-PFS at 2 years from registration will be reported.
Progression-free Survival (PFS) | Up to 5 years
  The PFS is defined as the duration from registration to either radiographic progression, clinical progression or death, whichever occurs first.
Percentage of Participants with PFS | 3 years
  Percentage of participants with PFS at 3 years from registration will be reported.
Overall Survival (OS) | Up to 5 years
  The OS is defined as the duration from registration to any death.
Percentage of Participants with Overall Survival (OS) | 3 years
  Percentage of participants with OS at 3 years from registration will be reported.
Cancer Specific Survival (CSS) | Up to 5 years
  The CSS is defined as the duration from registration to prostate cancer (PC)-related death. The PC-related death will be determined by each physician's discretion.
Percentage of Participants with CSS | 3 years
  Percentage of participants with CSS at 3 years from registration will be reported.
Time to Symptomatic Skeletal Event (TTSSE) | Up to 5 years
  The TTSSE is defined as the duration from registration to any first symptomatic skeletal event (SSE). The SSE is defined as 1 of the following: symptomatic pathological fracture, spinal cord compression, palliative radiation to bone and surgery to bone.
Patient Health Questionnaire-9 (PHQ-9) Score | Up to 5 years
  The PHQ-9 is a multipurpose self-reported inventory used for screening, diagnosing, and measuring the severity of mental status or depression of the patient. It contains 2 weeks recall of information and scores each of the 9 Diagnostic and Statistical Manual of Mental Disorders (4th edition; DSM-IV) criteria as "0" (not at all) to "3" (nearly every day).
Functional Assessment of Cancer Therapy for Prostate Cancer (FACT-P) Questionnaire Score | Up to 5 years
  The FACT-P consists of the FACT-General (FACT-G) and a PC-specific subscale. The FACT-G (Version 4) contains a 27-item questionnaire and is composed of 4 dimensions of health-related quality of life (HRQoL): physical well-being, social/family well-being, emotional well-being, and functional well-being. The PC-specific subscale is composed of 12 items, which span the dimensions of sexual function, bowel/bladder function, and pain. Each item for FACT-G subscale and PC-specific subscale is rated on a 0 to 4 Likert type scale. Higher scores represent better QoL.
Montreal Cognitive Assessment (MoCA) Score | Up to 5 years
  The MoCA is a rapid screening instrument for mild cognitive dysfunction. It assesses different cognitive domains: attention and concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation. The total possible score is 30 points; a score of 26 or above is considered normal.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K., Japan Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (77):
- Japan (77):
  - Akita University Hospital, Akita
  - Juntendo University Hospital, Bunkyō City
  - Tokyo Medical and Dental University Hospital, Bunkyō City
  - Chiba University Hospital, Chiba
  - Chiba Cancer Center, Chiba
  - University of Yamanashi Hospital, Chūō
  - Hospital of the University of Occupational and Enviromental Health, Fukuoka
  - Kyushu University Hospital, Fukuoka
  - Fukushima Medical University Hospital, Fukushima
  - Gifu University Hospital, Gifu
  - Harasanshin Hospital, Hakata-Ku
  - Hamamatsu University Hospital, Hamamatsu
  - Saitama Medical University International Medical Center, Hidaka
  - Hirosaki University Hospital, Hirosaki
  - Hiroshima University Hospital, Hiroshima
  - Tokyo Dental College Ichikawa General Hospital, Ichikawa
  - Tokyo Medical University Ibaraki Medical Center, Inashiki
  - Teikyo University Hospital, Itabashi Ku
  - Kanazawa Medical University Hospital, Kahoku-District
  - University Hospital Kyoto Prefectural University of Medicine, Kamigyo
  - St Marianna University Hospital, Kanagawa
  - Kanazawa University Hospital, Kanazawa
  - Nara Medical University Hospital, Kashihara
  - Kimitsu Chuo Hospital, Kisarazu-shi
  - Kagawa University Hospital, Kita Gun
  - Kobe University Hospital, Kobe
  - Kobe City Medical Center General Hospital, Kobe
  - Kochi Medical School Hospital, Kochi
  - Dokkyo Medical University Saitama Medical Center, Koshigaya
  - National Hospital Organization Shikoku Cancer Center, Matsuyama
  - Kitasato University Hospital, Minamiku
  - University of Miyazaki Hospital, Miyazaki
  - Iwate Medical University Hospital, Morioka
  - Aichi Medical University Hospital, Nagakute
  - Nagasaki University Hospital, Nagasaki
  - Nagoya City University Hospital, Nagoya
  - University of the Ryukyus Hospital, Nakagami Gun
  - Tokyo Metropolitan Police Hospital, Nakano
  - Miyagi Cancer Center, Natori-shi
  - Niigata University Medical And Dental Hospital, Niigata
  - Okayama University Hospital, Okayama
  - Osaka International Cancer Institute, Osaka
  - Kindai University Hospital, Osaka Sayama Shi
  - Gunma Prefectural Cancer Center, Ōta-ku
  - Shiga University of Medical Science Hospital, Ōtsu
  - Japan Community Health Care Organization Saitama Medical Center, Saitama
  - Sapporo Medical University Hospital, Sapporo
  - Hokkaido University Hospital, Sapporo
  - Tohoku University Hospital, Sendai
  - Tohoku Medical And Pharmaceutical University Hospital, Sendai
  - Jichi Medical University Hospital, Shimotsuke
  - Showa University Hospital, Shinagawa City
  - Japan Community Health care Organization Tokyo Shinjuku Medical Center, Shinjuku-ku
  - Chutoen General Medical Center, Shizuoka
  - Osaka University Hospital, Suita-shi
  - Osaka Medical and Pharmaceutical University Hospital, Takatsuki
  - Tokushima University Hospital, Tokushima
  - The Jikei University Hospital, Tokyo
  - Toranomon Hospital, Tokyo
  - Nippon Medical School Hospital, Tokyo
  - The Cancer Institute Hospital of JFCR, Tokyo
  - Tokyo Medical University Hospital, Tokyo
  - Ehime University Hospital, Toon-shi
  - Toyama University Hospital, Toyama
  - Fujita Health University Hospital, Toyoake
  - Mie University Hospital, Tsu
  - University of Tsukuba Hospital, Tsukuba
  - Yamaguchi University Hospital, Ube
  - Wakayama Medical University Hospital, Wakayama
  - Yamagata University Hospital, Yamagata
  - Yokohama Rosai Hospital, Yokohama
  - Yokohama City University Medical Center, Yokohama
  - Yokohama City University Hospital, Yokohama
  - Yokosuka Kyosai Hospital, Yokosuka
  - Tottori University Hospital, Yonago
  - University of Fukui Hospital, Yoshida
  - Oita University Hospital, Yufu

IPD SHARING:
Plan to Share IPD: No